CLINICAL TRIAL: NCT06012838
Title: The Systematic Approach for Identification of Cause Among Out-of-hospital Cardiac Arrest Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 202207125RIND
Record Dates: First submitted 2023-08-08; First posted 2023-08-28 (Actual); Last update posted 2023-08-28 (Actual); Status verified 2023-08

CONDITIONS: Out-Of-Hospital Cardiac Arrest
Keywords: Non-traumatic Out-Of-Hospital Cardiac Arrest; training program
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- cause classification of OHCA protocol (Experimental): The cause classification of OHCA protocol was developed by an expert cardiac arrest committee. A lecture concerning the Utstein's template, the epidemiology of cardiac arrest and the CCCA protocol was addressed to the participants.
  Interventions: Behavioral: Cause classification of OHCA protocol

INTERVENTIONS:
Behavioral: Cause classification of OHCA protocol — training program with cause classification of OHCA protocol

SUMMARY:
The cause of cardiac arrest mostly determines outcomes of cardiac arrest survivors. Identifying and treating the cause of cardiac arrest constitute a critical part in post-arrest care. However, the pathophysiology of cardiac arrest often encompasses multiple organ systems. Thus, forming accurate diagnosis for each case presents a daunting challenge, especially for unexperienced physicians. This study aims to evaluate whether a standardized protocol would improve the diagnostic proficiency for out-of-hospital cardiac arrest (OHCA) patients.

Sixteen Emergency Medicine Residents from National Taiwan University Hospital participated in this study. The cause classification of OHCA (CCCA) protocol was developed by an expert cardiac arrest committee, and a lecture concerning the Utstein's template, the epidemiology of cardiac arrest and the CCCA protocol was addressed. Pre-/post-lecture questionnaires regarding self-assessed diagnostic certainty and knowledge of cardiac arrest were obtained and compared to evaluate participants' learning effectiveness. To validate the efficiency of protocol, medical records of 586 non-traumatic OHCA adults with successful resuscitation and ICU admission were reviewed retrospectively, and the OHCA cause of each patient was identified by the trained residents following CCCA protocol. The primary outcome was the diagnostic consistency between protocolized diagnosis, expert diagnosis and the discharge diagnosis

DETAILED DESCRIPTION:
To identify the classification of OHCA cause, the cause classification of OHCA (CCCA) protocol was established based on previous studies, expert physician's experience and questionnaire of young physicians.

Residents from emergency department of National Taiwan University Hospital participated the program and received the lecture concerning the Utstein's template, the epidemiology of cardiac arrest, interpretation of examinations, and the CCCA protocol. To evaluate the learning effect of the lecture, pre-lecture and post-lecture questionnaire were designed, which included the knowledge for OHCA classification, confidence for correct diagnosis during CPR and after return of spontaneous circulation (ROSC), and the mandatory examinations for cause identification. Confidence level more than 50% was recognized as sufficient to make proper cause identification. The enrolled residents were asked to review the medical records of 3 non-traumatic adult OHCA patients before lecture and identified the OHCA cause by their own without the assist of the CCCA protocol. After lecture, another 3 medical records were reviewed by the participants with the use of the CCAC protocol. The consistency of OHCA cause between young physicians were evaluated before and after lecture, respectively.

To validate the efficiency of the CCCA protocol, these trained residents further identified the arrest cause of 586 non-traumatic adult OHCA patients who survived to ICU admission from January 2015 to July 2021 in NTUH following the established protocol.

The primary outcome was the consistency of OHCA cause between protocolized diagnosis, expert diagnosis and the discharge diagnosis. The diagnosis made by young physicians with protocol defined as protocolized diagnosis. The expert physician is an experienced emergency physicians specialized in both emergency and critical care, who has reviewed the medical records without the assistance of the established CCCA protocol. Expert diagnosis was recognized as diagnosis identified by expert physician. The discharge diagnosis is the major diagnosis related to index cardiac arrest.

Categorical variables are presented as numbers (percentages) and evaluated by the Chi-Squared test. The continuous variables are presented as mean ± standard deviation. The Light's kappa was used to evaluate the consistency of OHCA classification. The value ≤ 0.40 indicates minimal agreement, while value ≥ 0.80 represent strong and almost perfect consistency16-17. The statistical significance was set at p <0.05. All statistical analyses were performed using Statistical Package for Social Sciences Statistics (version 21.0; IBM, Chicago, IL, USA).

ELIGIBILITY:
Inclusion Criteria:

* Residents of National Taiwan University Hospital

Exclusion Criteria:

* Visiting staffs of National Taiwan University Hospital

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2022-08-10 (Actual); Primary Completion 2022-11-10 (Actual); Study Completion 2022-11-10 (Actual)

PRIMARY OUTCOMES:
diagnostic consistency between protocolized diagnosis and the discharge diagnosis | 3 months
  The diagnosis made by young physicians with protocol defined as protocolized diagnosis. Expert diagnosis was recognized as diagnosis identified by expert physician. The expert physician is an experienced emergency physicians specialized in both emergency and critical care, who has reviewed the medical records without the assistance of the established CCCA protocol. The discharge diagnosis is the major diagnosis related to index cardiac arrest. The Light's kappa was used to evaluate the consistency of OHCA classification.
diagnostic consistency between protocolized diagnosis and the expert diagnosis | 3 months
  The diagnosis made by young physicians with protocol defined as protocolized diagnosis. Expert diagnosis was recognized as diagnosis identified by expert physician. The expert physician is an experienced emergency physicians specialized in both emergency and critical care, who has reviewed the medical records without the assistance of the established CCCA protocol. The discharge diagnosis is the major diagnosis related to index cardiac arrest. The Light's kappa was used to evaluate the consistency of OHCA classification.

SECONDARY OUTCOMES:
Portion of sufficient confidence to make proper OHCA cause identification | 2 months
  To evaluate the learning effect of the lecture, pre-lecture and post-lecture questionnaire were designed. Confidence level more than 50% was recognized as sufficient to make proper cause identification. Categorical variables are presented as numbers (percentages) and evaluated by the Chi-Squared test.
the accuracy rates on the classification test of OHCA cause before and after the lecture | baseline, 2 weeks
  To evaluate the learning effect of the lecture, pre-lecture and post-lecture questionnaire were designed. The knowledge for OHCA classification was evaluated by the accuracy rates on each questionnaires. Categorical variables are presented as numbers (percentages) and evaluated by the Chi-Squared test.
diagnostic consistency between participants before and after the lecture | baseline, 2 weeks
  To evaluate the learning effect of the lecture, pre-lecture and post-lecture questionnaire were designed. The enrolled residents were asked to review the medical records of 3 non-traumatic adult OHCA patients before lecture and identified the OHCA cause by their own without the assist of the CCCA protocol. After lecture, another 3 medical records were reviewed by the participants with the use of the CCAC protocol. The consistency of OHCA cause between young physicians were evaluated before and after lecture, respectively. The Light's kappa was used to evaluate the consistency of OHCA classification.

CONTACTS AND LOCATIONS:
Overall Officials: Min-Shan Tsai, MD, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei County, Taiwan